CLINICAL TRIAL: NCT00473343
Title: An Open Multicenter, Phase III Study of Photodynamic Therapy With Metvix® Cream 160 mg/g in Patients With "High Risk" Basal Cell Carcinoma
Brief Title: Metvix PDT in Participant With "High Risk" Basal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC T310/00
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2021-06

CONDITIONS: Basal Cell Carcinoma
Keywords: Photodynamic therapy (PDT); PDT with Metvix cream; "High risk" BCC; Basal Cell carcinoma; Histologically confirmed complete response
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metvix® PDT (Experimental): Participants with basal cell carcinoma (BCC) lesions were administered to photodynamic therapy (PDT) with Metvix® cream 160 milligrams per gram (mg/g) applied for three hours, followed by illumination using non-coherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of 70-200 milliwatt per centimeter square (mW/cm*2) up to 13 weeks.
  Interventions: Drug: Metvix® cream

INTERVENTIONS:
Drug: Metvix® cream
  Other Names: Methyl 5-aminolevulinate hydrochloride

SUMMARY:
Photodynamic therapy (PDT) is the selective destruction of abnormal cells through light activation of a photosensitiser in the presence of oxygen. These cells accumulate more photosensitiser than normal cells. The photosensitiser generates reactive oxygen species upon illumination.

For skin diseases, there has been an increasing interest in using precursors of the endogenous photoactive porphyrins. The most commonly used precursors have been 5-aminolevulinic acid (ALA) and its derivatives. The present test drug, Metvix®, contains the methyl ester of ALA, which penetrates the lesions well and shows high lesion selectivity .

BCC is a highly frequent skin malignancy, and accounts for approximately 75% of all non-melanoma skin cancers. It is the most common cancer in humans. Several non-pharmacological treatment modalities are used for BCC, including excision surgery, curettage and electrodesiccation, cryosurgery and more advanced modalities like radiation therapy, plastic surgery with reconstruction and Moh's surgery. The treatment used depends on the type, size, depth and localisation of the BCC lesion. Treatment options for BCC give good response rates in the majority of participants but are inadequate in a small group of participants defined as "high-risk" BCC.

In this particular participant group, even a moderate complete response rate with good cosmetic results may be considered beneficial, since the number of participant who have to receive more advanced therapy with the possibility of high morbidity and poor cosmetic outcome was reduced. Even a partial response is of clinical interest since the remaining tumour was require less extensive surgery. In the case of treatment failure, Metvix PDT does not interfere with the use of other treatment modalities.

The variable "complete response" after one or two Metvix treatment cycles was used as the basis for the justification of sample size.

DETAILED DESCRIPTION:
Prospective, open, multicenter study. The high risk BCC lesions were treated with Metvix cream. A biopsy confirming the diagnosis of each BCC lesion should have been taken within 6 months prior to treatment. The participants was receive one or two treatment cycles each consisting of two Metvix PDT treatments 7 days apart (Lesions that did not respond completely after three months received a second PDT treatment cycle).

The primary end-point was the histologically confirmed complete response rate within a participant (No BCC cells in the biopsy taken 3 months after the last treatment).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of BCC lesions verified by histology (2-3 mm punch biopsy)
* Males or females above 18 years of age.
* Written informed consent. AND

Participants with high risk of surgical complications due to:

* Anticoagulant medication or bleeding disorders
* Cardiac risk factors
* Anaesthetic contraindications
* Poor surgical compliance because of participant refusal, dementia, or inability to perform wound care.

OR

• Participants with "high-risk BCC lesion(s). A "high-risk" BCC lesion is defined as:

A large BCC lesion with the largest diameter:

* Equal to or greater than 15 mm on extremities, except below the knees, where largest diameter should be equal to or greater than 10 mm
* Equal to or greater than 20 mm on the trunk
* Equal to or greater than 15 mm in the face, or A lesion in the mid-face region (H-zone according to Swanson) or on the ear In participants with more then 6 eligible lesions, the 6 lesions to be treated was randomly chosen.

Exclusion Criteria:

* Prior treatment of the lesion within 4 weeks.
* A pure morpheaform and/or highly infiltrated lesion assessed clinically and/or by histology. A mixed nodular/morpheaform lesion which is not highly infiltrated (clinically) may be included.
* Participant with porphyria.
* Pigmented lesions.
* Known allergy to Metvix® or a similar compound.
* Participation in another clinical study either concurrently or within the last 30 days
* Participant with Gorlin's syndrome.
* Participant with Xeroderma pigmentosum
* Pregnant or breast-feeding (all women of child-bearing potential must document a negative pregnancy test and use contraception during the treatments and for at least one month thereafter).
* Conditions associated with a risk of poor protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2000-09 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Vinciullo, MD, Principal Investigator — Dermatology Surgery & Laser Centre, Perth
Locations (7):
- Australia (7):
  - Department of Dermatology, St. George Hospital, Kogarah, New South Wales
  - South East Dermatology, The Belmont Specialist Clinic, Carnia, Queensland
  - Department of Dermatology, Royal Adelaide Hospital, Adelaide, South Australia
  - Dermatology Department, The Queen Elisabeth Hospital, Adelaide, South Australia
  - Clinic B, Repatriation Campus, Austin & Repatriation Medical Centre, Heidelberg, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Dermatology Surgery & Laser Centre, The Perth Surgicentre, Perth, Western Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 102 participants were randomized at seven different center in Australia.
Period: Overall Study
Arm/Group | Metvix® PDT
Started | 102
Completed | 52
Not Completed | 50
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 8
Not completed — Treatment failure | 27
Not completed — Withdrew consent | 3
Not completed — Other un-specified reason | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment.
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 102
Age, Continuous [Mean (Full Range); unit: years] | 64 [26 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 102
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Histologically Confirmed Patient Complete Response (CR) 3 Months After Last Metvix PDT Cycle
Description: Patient Complete Response (CR) was defined as 100 percentage of the lesions within the participant having negative findings for nodular basal cell carcinoma (BCC) in the histological examination.
Time Frame: 3 months after last Metvix PDT cycle, up to 6 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 102
percentage of participants | 80

2. Secondary Outcome: Number of Lesion With Complete Response 3 Months After Last Metvix PDT Cycle
Description: Complete response was defined as no clinically visible BCC lesions in the treatment area.
Time Frame: 3 months after last Metvix PDT cycle, up to 6 months
Population: as for baseline characteristics
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 102
Number analyzed (lesions) | 165
lesions | 141

3. Secondary Outcome: Overall Cosmetic Outcome Assessed by Investigator 3 Months After the Last Metvix PDT Cycle
Description: Cosmetic outcome was assessed by both investigator and participants in participants with 100% of lesions in complete response. Overall cosmetic outcome was assessed with regard to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. The investigator graded the cosmetic outcome as:
  * excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared lo adjacent skin
  * good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin
  * fair: slight to moderate occurrence of scarring, atrophy or induration
  * poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: 3 months after the last metvix PDT cycle, up to 6 months
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment. Here overall "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 82
Participants
  Investigator: Excellent | 37
  Investigator: Good | 16
  Investigator: Fair | 28
  Investigator: Not applicable | 1

4. Secondary Outcome: Overall Cosmetic Outcome Assessed by Participants 3 Months After the Last Metvix PDT Cycle
Description: Cosmetic outcome was assessed by both investigator and participants in participants with 100% of lesions in complete response. Overall cosmetic outcome was assessed with regard to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. The participants graded the cosmetic outcome as:
  excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared lo adjacent skin good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin fair: slight to moderate occurrence of scarring, atrophy or induration poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: 3 months after the last metvix PDT cycle, up to 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 81
Participants
  Participants: Excellent | 40
  Participants: Good | 39
  Participants: Fair | 2
  Participants: Not applicable | 0

5. Secondary Outcome: Recurrence Rate in Complete Clearance Group
Description: Recurrence rate in complete clearance(CC) group was analyzed.
Time Frame: 12, 24, 36, 48 and 60 months after last Metvix PDT cycle, up to 5 years
Population: Intent-to-treat analysis set included all the participants enrolled in the study who received at least one dose of study treatment. Here overall "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. "Number analyzed", signifies those participants who were evaluable for this outcome measure at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 69
Participants
  12 months | 8
  24 months: number analyzed (Participants) | 57
  24 months | 16
  36 months: number analyzed (Participants) | 49
  36 months | 20
  48 months: number analyzed (Participants) | 46
  48 months | 21
  60 months: number analyzed (Participants) | 42
  60 months | 23

6. Secondary Outcome: Overall Cosmetic Outcome Assessed by Investigator 24, 36, 48, and 60 Months After the Last Metvix PDT Cycle
Description: Cosmetic outcome was assessed by both investigator and participants in participants with 100% of lesions in complete response. Overall cosmetic outcome was assessed with regard to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. The investigator graded the cosmetic outcome as:
  excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared lo adjacent skin good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin fair: slight to moderate occurrence of scarring, atrophy or induration poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: 24, 36, and 60 Months After the Last Metvix PDT Cycle, up to 5 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® PDT
Number analyzed (Participants) | 57
Participants
  Excellent: At 24 month | 34
  Good: At 24 month | 15
  Fair: At 24 month | 7
  Poor: At 24 month | 1
  Excellent: At 36 month: number analyzed (Participants) | 50
  Excellent: At 36 month | 31
  Good: At 36 month: number analyzed (Participants) | 50
  Good: At 36 month | 13
  Fair: At 36 month: number analyzed (Participants) | 50
  Fair: At 36 month | 6
  Excellent: At 60 month: number analyzed (Participants) | 43
  Excellent: At 60 month | 35
  Good: At 60 month: number analyzed (Participants) | 43
  Good: At 60 month | 7
  Fair: At 60 month: number analyzed (Participants) | 43
  Fair: At 60 month | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Month 60
Arm/Group | Metvix® PDT
All-Cause Mortality (participants affected / at risk) | 7/102
Serious Adverse Events (participants affected / at risk) | 10/102
Other Adverse Events (participants affected / at risk) | 88/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metvix® PDT (N=102)
Angina Pectoris (Cardiac disorders) | 1
Burning sensation skin (Skin and subcutaneous tissue disorders) | 1
Surgical intervention (General disorders) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stroke (Vascular disorders) | 1
Peripheral vascular disease (Vascular disorders) | 1
Systemic infection (Infections and infestations) | 1
Encephalopathy (Hepatobiliary disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metvix® PDT (N=102)
Pain (General disorders) | 3
Chest pain (General disorders) | 2
Influenza like symptom (General disorders) | 2
Back ache (General disorders) | 1
Leg pain (General disorders) | 1
Allergic reaction (Cardiac disorders) | 1
Cervical pain (General disorders) | 1
Heaviness in limbs (General disorders) | 1
Oedema peripheral (General disorders) | 1
Feeling cold (General disorders) | 1
Fatigue (General disorders) | 1
Sensation of warmth (General disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Stomach upset (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Basel cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Skin neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Infection (Infections and infestations) | 3
Infection fungal (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Herpes simplex (Immune system disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Pain neck shoulder (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Mental distress (Psychiatric disorders) | 1
psychosis (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Eye pain (Eye disorders) | 3
conjunctivitis (Eye disorders) | 1
Stroke (Vascular disorders) | 1
Skin warm (Vascular disorders) | 1
Peripheral vascular disease (Vascular disorders) | 1
Haematoma (Blood and lymphatic system disorders) | 1
Epistaxis (Blood and lymphatic system disorders) | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Application site reaction (General disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Surgical intervention (Surgical and medical procedures) | 9
Abrasion NOS (Surgical and medical procedures) | 1
Prostatic specific antigen INCR. (Surgical and medical procedures) | 1
Heart Failure (Cardiac disorders) | 1
Liver failure related to Chronic Hepatitis B infection (Hepatobiliary disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cerebrovascular accident (Vascular disorders) | 1
Metastatic squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes